CLINICAL TRIAL: NCT02810106
Title: Assessment of Myocardial Perfusion by Tomography and Scintigraphy in Patients With Cardiac Stress Test With Ischemia
Acronym: Perfusão
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PERFUSÃO
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2018-06

CONDITIONS: Myocardial Perfusion
Keywords: Spect; Stress Test; Myocardial Perfusion CT; CT angiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Cardiovascular diseases are important cause of death, and of these have highlighted the Coronary Artery Disease (CAD) and its various clinical manifestations. The chest pain suggestive of ischemic heart disease is frequent complaint in medical consultations and hospitalizations . Complementary tests and images exams for risk stratification as Cardiac Stress Test (ET), the Myocardial Perfusion scintigraphy of (SPECT) are established for risk stratification and assessment workup in suspected ischemic heart disease. Coronary tomography angiography (CTA) has emerged as a robust method for non-invasive assessment of CAD, showing data diagnostics that directly correlate with invasive coronary angiography. Recently, the Myocardial Perfusion by Tomography Computed (CTP) has emerged as a new technique to measure the flow limitation for coronary microcirculation. In clinical practice, the exercise testing with electrocardiogram changes compatible with myocardial ischemia can lead to other examinations for elucidation of ischemic etiology, the most usual myocardial scintigraphy. However, a SPECT without evidence of ischemia, does not explain ischemic electrocardiographic changes triggered by physical stress, although it is a good marker prognostic. A CTP is a emerging tool in the evaluation of myocardial ischemia. Recent studies point to a good accuracy of the method compared to nuclear medicine. To test this hypothesis, this study aims to evaluate whether the CTP has a better diagnostic performance in detecting of obstructive or not obstructive CAD compared to the SPECT in the population of patients with exercise stress testing compatible with myocardial ischemia, and the computed tomography angiography (CTA) as the reference method. In addition, data from the exercise test (functional capacity, hemodynamics, electrocardiogram changes) will be compared to findings of CTA and CTP.

DETAILED DESCRIPTION:
Patients will be recruited in private Nuclear Medicine Service to perform myocardial perfusion scintigraphy with physical stress (SPECT-ET) that present the exercise test (less than 60 days) positive for ischemia, as electrocardiographic criteria enshrined in current guidelines of the Brazilian Society of Cardiology. These patients will be invited to participate in the study, guided and included after signing an informed consent form.

Patients included in the study will be submitted to 2 images exams protocols:

1. Myocardial perfusion scintigraphy with physical stress (SPECT-ET):

   Patients referred from other services with exercise testing positive ischemic response will be instructed to discontinue the drugs in use that may affect the ET as negative and coronary vasodilator action inotropic drugs. They will undergo perfusion study myocardial scintigraphy (SPECT) at rest and physical stress (1 day protocol), starting with Sestamibi Tn in injection 99 mtc at a dose of 10 millicurie and capture resting scintigraphic images in Gamma Camera GE millenium. Then they will undergo phase of physical stress, with maximum ET exercise, until exhaustion or intense physical exertion on the Borg Scale modified under Bruce protocol. At the peak of the effort will be injected into the radio tracer TC-99m Sestamibi at a dose of 30 mCi (milli Curie), and then quantified in Gamma Camera GE millenium scintigraphic images after physical stress.

   During the exercise test electrocardiographic variables will be evaluated as magnitude and morphology of ST segment changes, precocity and duration of these changes, hemodynamic variables such as behavior of the pressure curve and clinical variables.

   The perfusion myocardial study by Gated SPECT (single-photon emission computed tomography) will be analyzed qualitatively by 2 experienced examiners and semi-quantitatively using severity scores widely validated in the literature (SSS - Summed Stress Score; SRS - Summed Rest Score: SDS - summed Difference Score).
2. Myocardial Perfusion and Angiography by Computed Tomography. Patients will undergo myocardial perfusion computed tomography with multiple detectors after dipyridamole, as established protocol anteriores10 studies, followed by coronary angiography at rest (CTA) in tomography with 128 multi-detector channels Optima 660 CT (GE ).

Patients will be instructed to perform absolute fast 4 hours for the exam, and fasting for 24 foods with caffeine and medications containing xanthine derivatives. It will be obtained venous access caliber in the right upper limb and cardiac monitoring continues. They will be assessed and recorded weight, height, blood pressure (BP), heart rate (HR) at rest and respiratory rate before, during and after the examination tomography.

The evaluation of the pharmacological stress PMTC be performed after dipyridamole administration in a dose of 0,56mg / kg for 4 minutes. images, according to protocol previously validated in this study instituição10 immediately after injection of iodinated contrast After 2 minutes of dipyridamole administration of completion will be performed. Approximately 60ml of nonionic iodinated intravenous contrast medium is administered by an automated gun to a 3ml / s.

After the stress phase and the pharmacological reversal with aminophylline (240 mg), will be held the control of heart rate (metoprolol 5 mg IV every 5 minutes [max. 20mg] with the objective of reaching a HR ≤ 60), for carrying out the acquisition of coronary angiography. The acquisition parameters for CTA (resting phase) will be individualized according to the weight, sex and heart rate of each patient, in order to maintain a total dose of not more radiation 15mSv therefore a safe dose of radiation with the image quality maintenance. three-dimensional reconstructions and perfusion algorithm will be performed with the use of dedicated workstation (ADW4.6 [GE]).

ELIGIBILITY:
Inclusion Criteria:

* Patients with positive exercise test for ischemia Age> 18 years

Exclusion Criteria:

* Creatinine above 1.5 mg / dL and urea above 50 mg / dl and / or creatinine clearance <than 60ml / kg / min
* Pregnant women
* Known patients allergic to iodinated contrast or dipyridamole
* COPD and asthma
* Systolic blood pressure < 100 mmHg
* Any other aspect that the researcher considers limiting the method

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers of the population with positive exercise test for ischemia
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
myocardial perfusion data | 2 years
  myocardial perfusion assessment by multidetector computed tomography in patients with ischemic exercise test

SECONDARY OUTCOMES:
Anatomical data | 2 years
  Evaluation of coronary anatomy by multidetector computed tomography in patients with ischemic exercise test

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Rodrigo Beraldo, Dr., Principal Investigator — Nuclear Medicine Service of Magsul and CT scan of Corpus Images; Tiago Augusto Magalhaes, PhD, Study Director — Department Resonance and Cardiac Tomography of the Heart Institute of the University of Sao Paulo; Carlos Eduardo Rochitte, Study Chair — Department Resonance and Cardiac Tomography of the Heart Institute of the University of Sao Paulo
Locations (1):
- Corpus Imagens, Pouso Alegre, Minas Geral, Brazil

IPD SHARING:
Plan to Share IPD: No